CLINICAL TRIAL: NCT04376840
Title: Prevalence of Long-term Respiratory Complications of Severe SARS-CoV-2 Pneumonia
Brief Title: Prevalence of Long-term Respiratory Complications of Severe SARS-CoV-2 Pneumonia - COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO20066
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-09

CONDITIONS: Severe SARS-CoV2 Pneumonia
Keywords: SARS-CoV2; long term; complication; pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults with severe SARS-CoV2 pneumonia (Experimental): adult with severe SARS-CoV2 pneumonia
  Interventions: Other: Blood sample and data record

INTERVENTIONS:
Other: Blood sample and data record — Blood sample and data record

SUMMARY:
Studies performed after coronavirus epidemics (severe acute respiratory syndrome coronavirus, SARS-CoV and Middle East respiratory syndrome coronavirus, MERS-CoV) have shown a long-term impact on respiratory morbidity, musculoskeletal and psycho-social repercussions.

Patients with SARS-CoV pneumonia had fibrotic pulmonary sequelae at 45 days (lower DLCO in 27.3% of cases and radiological lesions in 21.5% of cases). In the MERS-CoV pneumonia study, patients had radiological sequelae in 33% of cases and the 12-month evaluation showed persistence of radiological abnormalities in 23.7% of the cases despite an improvement in respiratory function.

Clinical presentation and therapeutic management of severe SARS-CoV-2 infection are in part similar to those induced by SARS-CoV and MERS-CoV. Long-term respiratory complications are therefore expected.

DETAILED DESCRIPTION:
Objective is to evaluate prevalence of long-term respiratory complications after severe SARS-CoV2 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with with severe SARS-CoV2 pneumonia
* Patient consenting to participate to the study
* Patient enrolled in the national healthcare insurance program

Exclusion Criteria:

* Patient under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
medium-term respiratory complications | 3 months
  Interstitial lung disease diagnosed with a thoracic CT-scan

SECONDARY OUTCOMES:
long-term respiratory complications | 12 months
  Interstitial lung disease diagnosed with a thoracic CT-scan

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Result] Perotin JM, Gierski F, Bolko L, Dury S, Barriere S, Launois C, Dewolf M, Chouabe S, Bongrain E, Picard D, Tran E, N'Guyen Y, Mourvillier B, Servettaz A, Rapin A, Marcus C, Lebargy F, Kaladjian A, Salmon JH, Deslee G. Cluster analysis unveils a severe persistent respiratory impairment phenotype 3-months after severe COVID-19. Respir Res. 2022 Aug 2;23(1):199. doi: 10.1186/s12931-022-02111-9. PMID 35918719